CLINICAL TRIAL: NCT04386486
Title: The Effect of BATHE Method on Preoperative Anxiety, Patient Satisfaction and Individual Anesthesia Concerns in Adults in Anesthesia Polyclinics
Brief Title: BATHE Method on Preoperative Anxiety, Patient Satisfaction and Individual Anesthesia Concerns
Acronym: BATHE Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University Hospital (Other)
Responsible Party: Principal Investigator, Ahmet Cemil Isbir, Assoc. Prof., Cumhuriyet University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: bathe-2019
Record Dates: First submitted 2020-05-09; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Anesthesia; Reaction; Anxiety Preoperative; Patient Satisfaction
Keywords: preoperative anxiety; anesthesia anxiety; BATHE method; APAIS; patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bathe group (Experimental): The patients were divided into two equal groups randomly first group is BATHE anamnesis group.
  Interventions: Other: Bathe anamnesis method
- standart anamnesis group (Sham Comparator): The patients were divided into two equal groups randomly second group is standart anamnesis group.
  Interventions: Other: standart anamnesis

INTERVENTIONS:
Other: Bathe anamnesis method — BATHE anamnesis (BA) is applied to first group and preoperative examinations are completed.
  Arms: bathe group
Other: standart anamnesis — standart anamnesis is applied to second group and preoperative examinations are completed.
  Arms: standart anamnesis group

SUMMARY:
In this study the goal is to determine the causes of concern among the patients who will undergo surgical operations and receive general anesthesia, to gauge their preoperative anxiety levels and to study the effects of the BATHE method on preoperative anxiety and patient satisfaction.

DETAILED DESCRIPTION:
In this study the goal is to determine the causes of concern among the patients who will undergo surgical operations and receive general anesthesia, to gauge their preoperative anxiety levels and to study the effects of the BATHE method on preoperative anxiety and patient satisfaction.

500 patients who were planned to undergo elective surgery and under general anesthesia as anesthesia method were included in the study. Demographic data of patients, their three biggest fears of anesthesia and APAIS scores were recorded. The patients were divided into two groups, they underwent BATHE anamnesis or standard anamnesis methods according to their groups, then their APAIS and patient satisfaction scores were recorded.

ELIGIBILITY:
Inclusion Criteria: A) ASA I-II patients

Exclusion Criteria:

A) ASA III-IV B) illiterate patients C) patients with known psychiatric disorders D) patients with chronic sedative E) antipsychotic drug use F) patients with a history of going to psychiatry in the last year G) patients with any cancer diagnosis were not included in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-02-10 (Actual)

PRIMARY OUTCOMES:
t-test | 0-30 minutes
  when measurements taken from two independent groups are compared, the independent T-test was used.

CONTACTS AND LOCATIONS:
Overall Officials: Cemil A Isbir, M.D., Study Director — Dr. at Cumhuriyet University Hospital
Locations (1):
- Cemil Ahmet Isbir, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share any data of any patients with other researchers.

REFERENCES:
- [Background] DeMaria S Jr, DeMaria AP, Silvay G, Flynn BC. Use of the BATHE method in the preanesthetic clinic visit. Anesth Analg. 2011 Nov;113(5):1020-6. doi: 10.1213/ANE.0b013e318229497b. Epub 2011 Aug 24. PMID 21865495